CLINICAL TRIAL: NCT01233661
Title: Short Atrioventricular Delay Pacing
Acronym: SAVD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 08060137
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2016-01

CONDITIONS: Chronically (i.e. Implanted for at Least Six Months) Dual-chamber Pacemaker; Stable Cardiac Status (i.e. no Hospitalizations or Cardiac Medication Changes Within 3 Months)
MeSH Terms: interventions — Lead

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- short AVD pacing (Experimental): short AVD pacing
  Interventions: Other: short AVD pacing ; prior (stable) programming
- prior (stable) programming (No Intervention): prior (stable) programming

INTERVENTIONS:
Other: short AVD pacing ; prior (stable) programming — short AVD pacing prior (stable) programming
  Arms: short AVD pacing

SUMMARY:
We intend to examine the effects of temporary elevation of atrial wall stress by shortening of the atrioventricular delay in patients with dual-chamber pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Chronically (i.e. implanted for at least six months) dual-chamber pacemaker
* Stable cardiac status (i.e. no hospitalizations or cardiac medication changes within 3 months)
* Ability to provide informed consent

Exclusion Criteria:

* Age <18 years or >80 years
* Pregnancy (if pregnancy is suspected, a urine pregnancy test will be performed)
* Recent (within 12 months) left ventricular ejection fraction <50%
* Significant valvular heart disease (mitral regurgitation of greater than mild severity, any degree of mitral stenosis, aortic stenosis or insufficiency of greater than mild severity)
* Prior coronary artery bypass graft or valve surgery, recent (i.e. within 3 months) acute coronary syndrome or percutaneous coronary intervention, or chronic stable angina
* History of clinically important atrial or ventricular tachyarrhythmias, defined as complex ventricular ectopy (i.e. couplets, triplets, or ventricular tachycardia), AF, atrial tachycardia, or other supraventricular tachycardias not cured with prior ablative therapy).
* Significant chronic systemic inflammatory or neoplastic disease
* Chronic renal or hepatic insufficiency. Renal insufficiency will be defined as a creatinine clearance of less than 20 cc/min. Evidence of hepatic insufficiency will consist of abnormal synthetic function (INR >1.4 without oral anticoagulant use, albumin < 3.0 mg/dL) or abnormal clearance function (total bilirubin >2.0).
* Uncorrected thyroid abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
serum biomarker concentrations | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — Universtity of Pittsburgh
Locations (1):
- Atrial Arrhythmia Center, UPMC, Pittsburgh, Pennsylvania, United States